CLINICAL TRIAL: NCT06190418
Title: Comparative Effects of Loaded and Unloaded Sit to Stand Strengthening Exercises on Functional Strength and Energy Expenditure in Children With Cerebral Palsy
Brief Title: Loaded Vs Unloaded Sit to Stand Strengthening Exercises in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0729
Record Dates: First submitted 2023-11-09; First posted 2024-01-05 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy,; Energy Expenditure,; Muscle Strength
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Loaded sit to stand strengthening exercise group (Active Comparator): This group will be provided with loaded sit to stand strengthening exercises in spastic diplegic children.1 repetition maximum of the load will be provided. Exercise will be conducted 3 times a week for 6 weeks, pre and post session functional strength of lower limb will be measured by performing functional strength tests and physiological cost index will be measured to calculate energy expenditure.
  Interventions: Other: Loaded sit to stand strengthening exercise
- Unloaded sit to stand strengthening exercise group (Active Comparator): This Group will be provided with unloaded sit to stand exercises in diplegic spastic CP, 3 times a week for 6 weeks. Pre and post session functional strength of lower limb muscles will be measured by performing functional strength tests and physiological cost index will be measured to determine energy expenditure.
  Interventions: Other: Unloaded sit to stand strengthening exercise

INTERVENTIONS:
Other: Loaded sit to stand strengthening exercise — This Group will be given with the wieghted vest equal to that of 1RM for each child and Sit-to-Stand Strengthening Excerise will be given 3 times per week for 6 weeks
  Arms: Loaded sit to stand strengthening exercise group
Other: Unloaded sit to stand strengthening exercise — This Group will be given with the Sit-to-Stand Strengthening Excerise without any external load for 3 times per week for 6 weeks
  Arms: Unloaded sit to stand strengthening exercise group

SUMMARY:
Cerebral palsy(CP) is non-progressive disorder, undergo mishap to the developing brain and it affect a person's ability to move and maintain balance and posture. Old name of CP is "Little's disease". Cerebral means having to do with the brain. Palsy means weakness or problems with using the muscles. In Spastic diplegic, muscle stiffness is mainly in the legs, with the arms less affected or not affected at all. The most common cause of spastic diplegia is Periventricular leukomalacia, more commonly known as neonatal asphyxia or infant hypoxia-a sudden in-womb shortage of oxygen-delivery through the umbilical cord. Strength exercise is any activity that makes your muscles work harder than usual.

The significance of this study is that it will define whether loaded or unloaded sit to stand strengthening exercises have good effect on muscle strength and energy expenditure in diaplegic CP. This will be a randomized clinical trial, data will be collected from District Head Quarter DHQ hafizabad. Study will be conducted on 32 patients. Inclusion criteria of this study is spastic diplegic CP children with age between 6 to 12 years, with GMFCS level 1 and 2 and those who are able to stand up from chair independently and maintain standing for more than 5 seconds without falling will be included.Diplegic CP children who had not received any strengthening exercise program in past 3 months and those less than 20 degrees limitation in passive range of motion in hip flexion will be included. Those diplegic spastic CP who have orthopedic intervention such as selective dorsal rhizotomy or botolinum toxin injection to lower extremities within past six months and orthopedic conditions or medical problems that prevented children from participating in exercises will be excluded. Group A will be provided with loaded sit to stand strengthening exercises. 1 repetition maximum(1-RM) will be used as loaded sit to stand test. Group B will be provided with unloaded sit to stand strengthening exercises. Pre and post session lower limb functional strength will be measured by performing functional strength tests while lower limb muscular strength will be measured via modified sphygmomanometer and physiological cost index will be measured to rule out energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Spastic diplegic cerebral palsy
* Age between 6 to 12 years
* Children with GMFCS level I and II
* Able to stand up from chair independently and maintain standing for more than 5 second without falling.
* Had not received any strengthening exercise program in past 3 months
* Parental commitment to allow participation without altering current activity

Exclusion Criteria:

* Participants with epileptic history and lower limb contractures are excluded
* Those who are unable to follow verbal command
* Have orthopedic intervention such as selective dorsal rhizotomy or botolinum toxin injection to lower extremities within past 6 months
* Orthopedic condition or medical problems that prevent children from participating in exercise

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Muscle Strength | Baseline and 6th week
  Muscle strength will be assessed by Bag method of Modified Sphygmomanometer
Energy Expenditure | Baseline and 6th week
  To find out energy expenditure, physiological cost index (PCI) will be measured. PCI will be calculated by using the following formula: PCI (beats/meter)= Final heart rate -Resting Heart Rate /speed of walking

SECONDARY OUTCOMES:
Functional Strenght -Lateral Step-up Test (on a 20 cm bench) | Baseline and 6th week
  To assess functional strength, following tests will be used:
  The Lateral Step-up Test (on a 20 cm bench)
Functional Strenght -Sit-to-Stand (from 90 flexion of the knee and hip to standing position) | Baseline and 6th week
  To assess functional strength, following tests will be used:
  The Sit-to-Stand (from 90 flexion of the knee and hip to standing position) Attain stand through half kneel, without using arms.

CONTACTS AND LOCATIONS:
Overall Officials: Wasifa Rauf, MSPT(Peads), Principal Investigator — Riphah International University
Locations (1):
- District Headquarter Hospital,, Hafizabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kusumoto Y, Nitta O, Takaki K. Impact of loaded sit-to-stand exercises at different speeds on the physiological cost of walking in children with spastic diplegia: A single-blind randomized clinical trial. Res Dev Disabil. 2016 Oct;57:85-91. doi: 10.1016/j.ridd.2016.06.006. Epub 2016 Jul 7. PMID 27394691
- [Background] Lee J, Suk MH, Yoo S, Kwon JY. Physical Activity Energy Expenditure Predicts Quality of Life in Ambulatory School-Age Children with Cerebral Palsy. J Clin Med. 2022 Jun 11;11(12):3362. doi: 10.3390/jcm11123362. PMID 35743433
- [Background] Liao HF, Liu YC, Liu WY, Lin YT. Effectiveness of loaded sit-to-stand resistance exercise for children with mild spastic diplegia: a randomized clinical trial. Arch Phys Med Rehabil. 2007 Jan;88(1):25-31. doi: 10.1016/j.apmr.2006.10.006. PMID 17207671